CLINICAL TRIAL: NCT00187980
Title: Sleep Disturbance in Lung Cancer Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Other Study IDs: CP 05-02
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The aim of this study is to 1-evaluate subjectively by questionnaires and objectively by ambulatory actigraphy the quality of sleep in patients with newly diagnosed lung cancer; 2- to correlate sleep quality index with quality of life, daytime alertness, Performans status and lung cancer staging at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed lung cancer age > 18 yrs Performans status < 3 Informed consent Life expectancy > 5 months

Exclusion Criteria:

Psychiatric disease Performans status > 2 Known sleep disorder

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Le Guen, Principal Investigator — University Hospital, Angers
Locations (1):
- UH, Angers, France